CLINICAL TRIAL: NCT04591639
Title: An Observational Cross-sectional Study and a Double-blind Placebo Controlled Randomised Controlled Trial to Assess the Effect of Dapagliflozin on Myocardial Calcium-handling in Patients With Heart Failure- The DAPA-MEMRI Trial.
Brief Title: The DAPA-MEMRI Trial
Acronym: DAPA-MEMRI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Edinburgh (Other)
Collaborators: AstraZeneca (Industry); NHS Lothian (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: AC20006
Record Dates: First submitted 2020-08-14; First posted 2020-10-19 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Heart Failure; Diabetic Cardiomyopathies
Keywords: Heart failure; Sodium glucose Co-transporter 2 inhibitor therapy; Manganese enhanced cardiac magnetic resonance imaging
MeSH Terms: conditions — Heart Failure; Diabetic Cardiomyopathies | interventions — dapagliflozin

STUDY DESIGN:
Intervention Model Description: The observational component of the study will have 4 cohort of participants (patients with type 2 diabetes without heart failure, patients with heart failure with or without diabetes and healthy volunteers) The randomised controlled trial component of the study will have 2 groups of patients - heart failure with or without type 2 diabetes
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: As above
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients with heart failure without type 2 diabetes (Other): 60 patients with heart failure without type 2 diabetes will be recruited and will either be randomised to placebo or Dapagliflozin after their baseline cardiac MRIs. They will have 2 cardiac MRIs (gadolinium and manganese enhanced) at baseline and further manganese enhanced cardiac MRI at 1 month post randomisation + gadolinium and manganese enhanced cardiac MRI at 6 months post randomisation.
  Interventions: Drug: Dapagliflozin 10 milligrams [Farxiga]; Drug: Placebo
- Patients with heart failure with type 2 diabetes (Other): 60 patients with heart failure with type 2 diabetes will be recruited and will either be randomised to placebo or Dapagliflozin after their baseline cardiac MRIs. They will have 2 cardiac MRIs (gadolinium and manganese enhanced) at baseline and further manganese enhanced cardiac MRI at 1 month post randomisation + gadolinium and manganese enhanced cardiac MRI at 6 months post randomisation.
  Interventions: Drug: Dapagliflozin 10 milligrams [Farxiga]; Drug: Placebo

INTERVENTIONS:
Drug: Dapagliflozin 10 milligrams [Farxiga] — Patients with heart failure with or without type 2 diabetes will be either randomised to 10mg Dapagliflozin once daily or matched placebo.
Drug: Placebo — Patients with heart failure with or without type 2 diabetes will be either randomised to 10mg Dapagliflozin once daily or matched placebo.

SUMMARY:
Diabetes mellitus is among the top 10 causes of death worldwide with an increasing incidence. Patients with diabetes are at risk of developing heart failure which is characterised by significant changes in the heart muscle including scarring and thickening. Contraction of the heart involves movement of calcium across the heart muscle and disruption of this process is an early change seen in heart failure. Recently, a drug therapy (SGLT2 inhibitor therapy) in patients with diabetes was shown to benefit patients with heart failure but the mechanisms of benefit are unknown.

Our hypothesis is that calcium handling is altered in patients with either type 2 diabetes mellitus (T2DM) or heart failure and that SGLT2 inhibitors can improve this in heart failure irrespective of the presence of T2DM.

Scanning the heart using magnetic resonance imaging (MRI) enables detailed assessment of its structure and function by using a new contrast 'dye' containing manganese that has shown advantages over traditional contrast. We plan to further test this new dye as it has the potential to track and quantify improvements in heart function over time and detect changes in calcium handling in the heart muscle, making it an ideal measure to identify the mechanisms of benefit from SGLT2 inhibitor therapy.

The study population will comprise patients with heart failure with and without type 2 diabetes, patients with type 2 diabetes without heart failure and healthy volunteers. Baseline comparisons will be made between the four groups before progressing to the randomised controlled trial with heart failure patients only. Patients will have a clinical assessment and blood tests, electrocardiogram, echocardiogram and MRI of the heart at each visit.

If successful, this study will give us significant insights into mechanisms of action of SGLT2 inhibitors in heart failure and will enable us to tailor specific treatments in heart failure patients.

DETAILED DESCRIPTION:
The study is designed to investigate the myocardial calcium handling in patients with heart failure with or without type 2 diabetes mellitus and if Dapagliflozin (study drug) improves the myocardial calcium handling in patients with heart failure and diabetes mellitus.

We propose to conduct this study in two parts.

1. OBSERVATIONAL CROSS-SECTIONAL STUDY

   An observational cross-sectional study will be undertaken to compare myocardial calcium in patients with diabetes mellitus and normal left ventricular ejection fraction (n=20), patients with heart failure in the absence of diabetes mellitus (n=60), and patients with both diabetes mellitus and heart failure (n=60). They will be compared with healthy volunteers (n=20).

   There will be an initial meeting, where informed consent will be documented and a medical assessment including blood tests will be undertaken as well as an echocardiogram will be performed. Healthy volunteers will only undergo Manganese enhanced cardiac MRI scan. The other cohorts will undergo a gadolinium enhanced cardiac MRI scan on their first visit. On a subsequent visit, they will undergo 1 cardiac Manganese enhanced Manganese MRI scan (MEMRI) which lasts 45-60 minutes. Participants will be monitored with blood pressure and ECG monitoring throughout the MEMRI scan. Patients will be offered an anti-sickness medication if required following the MEMRI scan.
2. RANDOMISED CONTROLLED TRIAL

We will undertake a randomised double-blind placebo controlled trial of patients with heart failure with (n=60) and without (n=60) type 2 diabetes mellitus. These participants would have been recruited as part of the observational study as described above from out-patient clinics at the Edinburgh Heart Centre. If all eligibility criteria are met, patients will be randomised to receive treatment with either Dapagliflozin 10 mg, or matched placebo, once daily for 6 months at a ratio of 1:1. Detailed clinical assessment including history and examination, blood sampling, electrocardiogram, echocardiogram and cardiac MRI will be collected at baseline, 1 and 6 months.

There will also be a 3 month safety visit after randomisation to record any adverse events.

ELIGIBILITY:
Inclusion Criteria:

Patients with heart failure (with or without type 2 diabetes mellitus)

* Aged over 18 years
* Diagnosis of symptomatic reduced ejection fraction heart failure for at least 2 months
* Left ventricular ejection fraction ≤40%
* Elevated N-terminal pro B-type natriuretic peptide (>125 pg/mL)
* Clinical diagnosis of type 2 diabetes mellitus for 50% of patient population - on stable therapy for at least 12 months or more.

Patients with Type 2 Diabetes Mellitus and no heart failure

* Aged over 18 years
* Clinical diagnosis of type 2 diabetes mellitus (diagnosed by either HbA1c of 48mmol/mol (6.5%) or greater or fasting plasma glucose level of 7mmol/L or greater at the time of diagnosis)

  - on stable therapy for at least 12 months or more.
* Normal left ventricular systolic ejection fraction

Healthy Volunteers

* Aged over 18 years
* Normal left ventricular ejection fraction and glycaemia
* No clinically significant co-morbid conditions

Exclusion Criteria:

Patients with heart failure (with or without type 2 diabetes mellitus)

* Receiving an SGLT2 inhibitor within 8 weeks of enrolment
* Previous intolerance of, or contraindication to, an SGLT2 inhibitor
* Standard magnetic resonance imaging safety exclusions
* Severe renal impairment (eGFR <30millilitre/min. 1.73m2)
* Type 1 diabetes mellitus
* Symptomatic hypotension or systolic blood pressure <95 mmHg
* Recent (within 12 weeks) hospitalisation for heart failure, acute cardiovascular event (such as myocardial infarction or stroke) or coronary re-vascularisation.
* 2nd or 3rd degree atrioventricular block Atrial fibrillation or flutter with poor ventricular rate control (>100 /min)
* Heart failure due to restrictive cardiomyopathy, active myocarditis, constrictive pericarditis, hypertrophic (obstructive) cardiomyopathy or uncorrected primary valvular disease
* New York Heart Association grade IV heart failure
* Obstructive liver function testing abnormalities
* Concomitant digoxin, diltiazem or verapamil therapy.

Patients with type 2 diabetes mellitus and no heart failure

* Other major clinically significant co-morbid conditions
* History of ischaemic heart disease or present history suggestive of probable clinically significant underlying ischaemic heart disease
* Standard magnetic resonance imaging safety exclusions
* Moderate or severe renal impairment (eGFR <45 mL/min. 1.73m2)
* Receiving a SGLT2 inhibitor at any time
* Symptomatic hypotension or systolic blood pressure <95 mmHg
* Abnormal electrocardiogram
* Clinically significant abnormalities of clinical haematology or biochemistry measurements.

Healthy Volunteers

* Major or clinically significant cardiovascular disease
* Diabetes mellitus
* Receiving an SGLT2 inhibitor at any time
* Standard magnetic resonance imaging safety exclusions
* Moderate or severe renal impairment (eGFR <45 mL/min. 1.73m2)
* Symptomatic hypotension or systolic blood pressure <95 mmHg
* Abnormal electrocardiogram
* Clinically significant abnormalities of clinical haematology or biochemistry measurements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2020-08-19 (Actual); Primary Completion 2028-07-28 (Estimated); Study Completion 2028-07-28 (Estimated)

PRIMARY OUTCOMES:
Rate of change in myocardial T1 values with manganese enhanced cardiac MRI | 6 months

SECONDARY OUTCOMES:
Left ventricular ejection fraction measured in percentage on cardiac MRI | 6 months
Left ventricular mass measured in grams on cardiac MRI | 6 months
Cardiac biomarkers like N-terminal pro B-type natriuretic peptide in nanogram per litre | 6 months
Markers of diabetes control including glucose in millimoles per litre | 6 months
Clinical measures such as heart rate in beats per minute | 6 months
Extracellular volume in percentage as per cardiac MRI measurements | 6 months
Global longitudinal strain in percentage as calculated on cardiac MRI | 6 months
Clinical measures such as body weight in Kilograms | 6 months
Clinical measures such as blood pressure in millimetres of mercury | 6 months
Cardiac biomarkers like high sensitivity cardiac troponin I in nanogram per litre | 6 months
Measures of glucose control like glycated haemoglobin (HbA1c) in millimoles per mole | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- University of Edinburgh, Edinburgh, Scotland, United Kingdom

IPD SHARING:
Plan to Share IPD: No